CLINICAL TRIAL: NCT04113980
Title: Effects of Distraction Methods on Pain Perceptions and Anxiety Levels in Children During the Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Tuba Koc Ozkan, Principal Investigator, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Adiyaman University/2018/2-23
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Acute Pain; Nursing Caries
Keywords: acute pain; anxiety; children; blood collection; nursing
MeSH Terms: conditions — Acute Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- music group (Experimental): The children in the groups were distracted by listening music 2 minutes before venipuncture, until the process was over.
  Interventions: Other: music group
- kaleidescope group (Experimental): The children in the groups were distracted by kaleidoscope 2 minutes before the blood collection, until the process was over.
  Interventions: Other: kaleidoscope group
- video group (Experimental): The children in the groups were distracted by watching cartoon 2 minutes before the blood collection, until the process was over.
  Interventions: Other: video group
- control group (No Intervention): No intervention was made to children in the control group

INTERVENTIONS:
Other: music group — The children in the groups were distracted by music 2 minutes before venipuncture, until the process was over
  Arms: music group
Other: kaleidoscope group — The children in the groups were distracted by kaleidoscope 2 minutes before venipuncture, until the process was over
  Arms: kaleidescope group
Other: video group — The children in the groups were distracted by watching video 2 minutes before venipuncture, until the process was over
  Arms: video group

SUMMARY:
Aim:This study was conducted to investigate the effects of music, kaleidoscope and video watching methods on children's pain perception and anxiety level during the blood collection procedures.

Methods: This randomized controlled experimental study was carried out with 134 children in the 5-10 age group in the pediatric blood collection unit of a Training and Research Hospital between August and November 2018. In the study, nonpharmacological methods were applied to the children in the experimental groups (Music Group (n=33), Kaleidoscope Group (n=36), Video Group (n=31). The routine blood collection procedure was used for the children in the control group (n=34). The data were collected using the "Introductory Information Form", "Children's Fear and Anxiety Scale (CFAS)", and the "Wong-Baker Faces Pain Rating Scale (WB-FPRS)".

ELIGIBILITY:
Inclusion Criteria:

* being healthy
* ability to express himself/herself verbally
* no analgesic taken in the last 6 hours
* having no visual or auditory problems

Exclusion Criteria:

* chronic disease
* mental disease
* neurological disease

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Children Fear Scale | 1 minute
  The Children Fear Scale was used to evaluate the children's fear and anxiety. Children Fear Scale is a 0-4 scale, showing five faces that range from a neutral expression (0 = no anxiety) to a frightened face (4 = severe anxiety). Preprocedural and procedural pain, and anxiety were evaluated
Wong Baker Face Pain Scale | 1 minute
  The Wong Baker Faces scale is a 0-10 scale. Six faces on the cards show a range of emotions from a smiling face (0 very happy/no pain) to a crying face (10 'hurts worst').

CONTACTS AND LOCATIONS:
Locations (1):
- Adiyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No